CLINICAL TRIAL: NCT06880432
Title: Sarcopenic Obesity: Estimation of Prevalence and Identification of Clinical and Biological Determinants in a Cohort of Adult Obese Patients and Longitudinal Follow-up
Acronym: OBESAR-2
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: RBHP 2024 BOIRIE
Record Dates: First submitted 2025-03-05; First posted 2025-03-17 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Obesity and Overweight
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cohort (Other): Collection of clinical and paraclinical data (biological and anthropometric) for evaluation of sarcopenic obesity in obese patients.
  Interventions: Other: Collection of fluid samples

INTERVENTIONS:
Other: Collection of fluid samples — - Blood sampling, urine sampling and tissue sampling

SUMMARY:
Context: Obesity, defined as excessive body fat, can lead to disability and loss of autonomy. If there is concomitant quantitative and qualitative muscle loss, sarcopenic obesity (SO) is suspected in this context. Although this clinical entity was defined several years ago, it is only very recently that precise assessment criteria have been established for screening and diagnosing this pathology (Donini et al. 2022).

Defined by the ESPEN/EASO consensus, SO has various consequences for health, particularly in terms of mobility and worsening of co-morbidities. It is therefore necessary to screen for SO, to determine its prevalence in the general population and to identify the determining factors in the loss of muscle mass during obesity. Most studies on the prevalence of sarcopenic obesity focus on the elderly population, bearing in mind that the prevalence of this syndrome in the elderly will increase rapidly as a result of the shift in the incidence of obesity from adults to this population in the coming decades.

The aim of this project is to determine the prevalence and determining or predisposing factors for sarcopenic obesity in a population of obese people in a broad age range (18-70 years).

Longitudinal follow-up of this cohort is planned in order to assess multifactorial changes (body composition, muscle function and physical performance) at 5 and 10 years after their inclusion in the OBESAR-2 study. In addition, patients who have undergone bariatric surgery will also be followed in the shorter term to analyse the phenotypic changes induced by rapid weight loss on muscle loss.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-70
* Sex: men and women
* Clinical nutrition patient receiving a metabolic assessment to optimise clinical and paraclinical management
* Patient meeting obesity criteria defined by BMI > 30 kg/m².
* Patient of legal age who has given free, informed and signed consent
* Patient covered by social security

Non-inclusion criteria :

* Patients with cancer or severe chronic disease (renal failure, respiratory failure, liver failure)
* Patients with neuromuscular disease
* Patient with total walking disability
* Patients who are minors
* Patient refusing to take part in the study
* Pregnant or breast-feeding women
* Under guardianship, curatorship, deprived of liberty or under court protection
* Patient who has taken part in the OBESAR study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2039-12 (Estimated); Study Completion 2039-12 (Estimated)

PRIMARY OUTCOMES:
To estimate the prevalence of sarcopenia in a population of adult subjects with obesity, at baseline and at 5 and 10 years. | Day 1 / 5 years /10 years
  The primary endpoint is the presence of sarcopenic obesity at inclusion, 5 years and 10 years post-inclusion, assessed according to the latest current recommendations, i.e. impaired muscle function and impaired body composition (Donini et al. 2022).
  A patient presents with sarcopenic obesity when there is an alteration in muscle function AND an alteration in body composition.
  For impaired muscular function, strength measured with the handgrip is considered pathological when it is less than 27kg for men and less than 16kg for women.
  Altered body composition is considered to exist when fat mass is greater than 39, 41 and 43% for women aged between 20 and 39, 40 and 59, and 60 and 79 respectively, and greater than 26, 29 and 31% for men aged between 20 and 39, 40 and 59, and 60 and 79 respectively, AND SMM/W (Skeletal Muscle Mass/Weight) is less than 37% in men and 27.6% in women.

SECONDARY OUTCOMES:
% of patients with the factors associated with sarcopenia | Day 1 / 5 years /10 years
  Study the factors associated with sarcopenia by considering the clinical and biological characteristics of obese patients.
concentration of biomarkers in a group of obese patients with sarcopenia using the biobank. | Day 1 / 5 years /10 years
  Identify plasma, serum, genetic and urinary biomarkers in a group of obese patients with sarcopenia using the biobank.
Evaluate the degree of severity of sarcopenic obesity over time using the ESPEN/EASO consensus staging system. | Day 1 / 5 years /10 years
% change of parameters measured to identify the group at risk of accelerated decline | 5 years /10 years
  Evaluate 5- and 10-year trends in anthropometric measurements, muscle function, metabolic parameters and body composition to estimate the group at risk of accelerated decline
% of evolution of biomarkers | Day 1 / 5 years /10 years
  Evaluate changes in plasma, serum, genetic and urinary biomarkers in the same population 5 and 10 years after the inclusion visit, and assess the relationship between changes in biomarkers and changes in sarcopenia using the biobank.
% of risk of various health problems (diabetes, hypertension, etc.) between sarcopenic and non-sarcopenic patients. | Day 1 / 5 years /10 years
  Study the risk of various health problems (diabetes, hypertension, etc.) between sarcopenic and non-sarcopenic patients.
% of patients with the factors associated with sarcopenia in the subgroup of patients undergoing bariatric surgery. | Day 1 /Day of surgery/ 6 months after surgery/ 12 months after surgery/ 5 years /10 years]
  Study the factors associated with sarcopenia by considering the clinical and biological characteristics of obese patients.
concentration of biomarkers in a group of obese patients with sarcopenia using the biobank in the subgroup of patients undergoing bariatric surgery. | Day 1 /Day of surgery/ 6 months after surgery/ 12 months after surgery/ 5 years /10 years]
  Identify plasma, serum, genetic and urinary biomarkers in a group of obese patients with sarcopenia using the biobank.
Evaluate the degree of severity of sarcopenic obesity over time using the ESPEN/EASO consensus staging system in the subgroup of patients undergoing bariatric surgery. | Day 1 /Day of surgery/ 6 months after surgery/ 12 months after surgery/ 5 years /10 years]
% of evolution of biomarkers in the subgroup of patients undergoing bariatric surgery. | Day 1 /Day of surgery/ 6 months after surgery/ 12 months after surgery/ 5 years /10 years
  Evaluate changes in plasma, serum, genetic and urinary biomarkers in the same population 5 and 10 years after the inclusion visit, and assess the relationship between changes in biomarkers and changes in sarcopenia using the biobank.
% of risk of various health problems (diabetes, hypertension, etc.) between sarcopenic and non-sarcopenic patients in the subgroup of patients undergoing bariatric surgery. | Day 1 /Day of surgery/ 6 months after surgery/ 12 months after surgery/ 5 years /10 years]
  Study the risk of various health problems (diabetes, hypertension, etc.) between sarcopenic and non-sarcopenic patients.

CONTACTS AND LOCATIONS:
Overall Officials: Yves BOIRIE, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France